CLINICAL TRIAL: NCT00428818
Title: Empiric Therapy With Trimethoprim-Sulfamethoxazole or Doxycycline for Outpatient Skin and Soft Tissue Infections in an Area of High MRSA Prevalence: A Prospective Randomized Trial
Brief Title: Trimethoprim-Sulfamethoxazole or Doxycycline for Skin and Soft Tissue Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 072005-011
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2007-01-30 (Estimated); Status verified 2007-01

CONDITIONS: Infection
Keywords: MRSA
MeSH Terms: conditions — Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Doxycycline

INTERVENTIONS:
Drug: trimethoprim-sulfamethoxazole or doxycycline

SUMMARY:
Background: In many communities, skin and soft tissue infections (SSTI) with MRSA have become more prevalent than infections with β-lactam susceptible bacteria. This has necessitated altered empiric antimicrobial therapy of SSTI to cover MRSA.

Objective: To evaluate empiric therapy with trimethoprim-sulfamethoxazole or doxycycline for outpatient SSTI in an area of high MRSA prevalence.

Design: Randomized, prospective, open-label investigation. Setting: Emergency Department of Parkland Hospital in Dallas, Texas. Patients: Adults with SSTI. Intervention: Empiric oral therapy with trimethoprim-sulfamethoxazole (160 mg/800 mg, twice daily) or doxycycline (100 mg, twice daily).

Measurement: The primary endpoint was clinical failure defined as hospitalization or change in antibiotic therapy over the 10 to 14 days after initial emergency department evaluation.

DETAILED DESCRIPTION:
As MRSA in more likely to be isolated from a SSTI than is a β-lactam susceptible organism at Parkland Hospital in Dallas, Texas, we performed a randomized, prospective, open-label investigation in our emergency department to determine the efficacy of empiric therapy using off-patent oral antibiotics (trimethoprim-sulfamethoxazole 160 mg/800 mg twice daily or doxycycline 100 mg twice daily for 7 days) for the outpatient treatment of SSTI abscesses, requiring wound packing after incision and drainage but not requiring hospitalization. Only SSTI requiring wound packing were enrolled to eliminate the inclusion of smaller SSTI not requiring wound packing.

This investigation was approved by The University of Texas Southwestern Medical Center Institutional Review Board and included adults (≥ 18 years old) who were willing and able to provide informed consent. Inclusion criteria included being able to return for follow-up at 2 to 5 days after enrollment and being accessible by telephone for follow-up assessment at 10 to 14 days and 28 to 35 days after enrollment. Exclusion criteria excluded patients with contraindications or history of hypersensitivity reaction to any of the study treatment regimens, an infected prosthesis or device, concomitant bacteremia or deep infections (e.g. osteomyelitis, necrotizing fasciitis, endocarditis), diabetic foot infections, known immunodeficiency, pregnant or breastfeeding, requirement of additional antimicrobial agents, and those who did not obtain assigned antibiotics.

The primary endpoint of this study was clinical failure defined as subsequent hospital admission, administration of intravenous antibiotics, or change in oral antibiotics over a period of 10-14 days after initial emergency department presentation. Repeated outpatient incision and drainage of the SSTI at 2 to 5 days after enrollment was not considered a clinical failure, if antibiotics were not changed and intravenous antibiotics were not administered. The trial enrolled patients from October 2005 to May 2006. Method of randomization was by generation of random numbers using www.randomizer.org, and alternately assigning these to the two treatment groups, and then sorting the numbers consecutively to determine the sequence of assigning treatment group to consecutively recruited patients. Statistical analysis was performed with SigmaStat 3.0 software (SPSS Inc., Chicago, Illinois). This investigation had no external funding.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient treatment of SSTI abscesses, requiring wound packing after incision and drainage but not requiring hospitalization.
* Adults (≥ 18 years old) who were willing and able to provide informed consent.
* Able to return for follow-up at 2 to 5 days after enrollment and being accessible by telephone for follow-up assessment at 10 to 14 days and 28 to 35 days after enrollment.

Exclusion Criteria:

* Exclusion criteria excluded patients with contraindications or history of hypersensitivity reaction to any of the study treatment regimens, an infected prosthesis or device, concomitant bacteremia or deep infections (e.g. osteomyelitis, necrotizing fasciitis, endocarditis), diabetic foot infections, known immunodeficiency, pregnant or breastfeeding, requirement of additional antimicrobial agents, and those who did not obtain assigned antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2005-08; Study Completion 2006-07

PRIMARY OUTCOMES:
The primary endpoint was clinical failure defined as hospitalization or change in antibiotic therapy over the 10 to 14 days after initial emergency department evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Hardy, MD, Study Director — University of Texas Southwestern Medical Center